CLINICAL TRIAL: NCT02007720
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled Phase III Study to Evaluate the Efficacy, Safety and Tolerability of Serelaxin When Added to Standard Therapy in Acute Heart Failure Patients
Brief Title: Efficacy, Safety and Tolerability of Sexelaxin When Added to Standard Therapy in AHF
Acronym: RELAX-AHF-ASIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated based on results from pivotal adult AHF study CRLX030A2301
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A2302
Record Dates: First submitted 2013-11-20; First posted 2013-12-11 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Acute Heart Failure
Keywords: Serelaxin,; WHF,; Likert Scale,; RELAX-AHF-ASIA,; RLX030,; AHF,; acute heart failure
MeSH Terms: interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive continuous intravenous infusion of matching placebo serelaxin for 48 hours.
  Interventions: Drug: Placebo; Other: Standard of CareTherapy
- Serelaxin (Experimental): Patients will receive continuous intravenous infusion of serelaxin(30 µg/kg/day) for 48 hours.
  Interventions: Drug: Serelaxin; Other: Standard of CareTherapy

INTERVENTIONS:
Drug: Serelaxin — Intravenous infusion
  Arms: Serelaxin
Drug: Placebo — Intravenous infusion
  Arms: Placebo
Other: Standard of CareTherapy — This treatment can include but is not limited to intravenous and/or oral diuretics, ACE inhibitors/angiotensin receptor antagonists, β blockers, and aldosterone receptor antagonists, etc.

SUMMARY:
The purpose of the study was to evaluate the efficacy, safety and tolerability of intravenous infusion of serelaxin, when added to standard therapy, in acute heart failure (AHF) patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age, with body weight ≤160 kg
* Hospitalized for AHF; AHF is defined as including all of the following measured at any time between presentation (including the emergency department and outpatient clinic) and at the end of screening:

  * Persistent dyspnea at rest or with minimal exertion at screening and at the time of randomization
  * Pulmonary congestion on chest radiograph
  * Brain natriuretic peptide (BNP) ≥500 pg/mL or NT-proBNP ≥2,000 pg/mL
* Systolic BP ≥125 mmHg at the start and at the end of screening
* Able to be randomized within 16 hours from presentation to the hospital, including the emergency department and outpatient clinic
* Received intravenous furosemide of at least 40 mg total (or equivalent) at any time between presentation (this includes outpatient clinic, ambulance, or hospital including emergency department) and the start of screening for the study for the treatment of the current acute HF episode
* Renal impairment defined as an estimate glomerular filtration rate using the between presentation and randomization of ≥ 25 and ≤75mL/min/1.73m2, calculated using the Modification of Diet in Renal Disease formula (or modified sMDRD formula according to specific ethnic groups and local practice guidelines).

Exclusion Criteria:

* Dyspnea primarily due to non-cardiac causes
* Temperature >38.5°C (oral or equivalent), sepsis, active and clinically significant infection requiring IV anti-microbial treatment or known presence or evidence of Human Immunodeficiency Virus (HIV) infection (based on history and/or clinical findings, including laboratory results obtained during screening period).
* Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrollment

  *Patients with systolic blood pressure >180 mmHg at the end of screening
* AHF due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate <45 beats per minute, or atrial fibrillation/flutter with sustained ventricular response of >130 beats per minute
* Hepatic disease unrelated to Heart Failure etiology and as determined by any one of the following: AST and/or ALT values exceeding 3 X ULN and/or bilirubin > 1.5 X ULN at screening or history of hepatic encephalopathy, esophageal varices, or portacaval shunt, or a diagnosis of cirrhosis by any means, or evidence of chronic Hepatitis B (presence of hepatitis B surface antigen production: positive HBsAg), or chronic Hepatitis C infection (presence of Hepatitis C genetic replication: positive Hepatitis C viral RNA, based on history and/or clinical findings, including laboratory results obtained during screening period).

  *Significant uncorrected left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area <1.0 cm2 or mean gradient >50 mmHg on prior or current echocardiogram), and severe mitral stenosis
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past year with a life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (108):
- China (15):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Yangzhou, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Zhujing, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- India (7):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Rajasthan, India
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
- Japan (46):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Kamogawa, Chiba
  - Novartis Investigative Site, Saijō, Ehime
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Kushiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kan’onjichō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Yatsushiro, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Uji, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nakano, Nagano
  - Novartis Investigative Site, Saku, Nagano
  - Novartis Investigative Site, Ueda, Nagano
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Wako, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Kakegawa, Shizuoka
  - Novartis Investigative Site, Akishima, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Tanabe, Wakayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
- Jordan (2):
  - Novartis Investigative Site, Amman, JOR
  - Novartis Investigative Site, Amman
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Hazmiyeh
- Malaysia (6):
  - Novartis Investigative Site, Kuala Lumpur, MYS
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur, Selangor
  - Novartis Investigative Site, Sungai Buloh, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Philippines (7):
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, San Juan City
- Novartis Investigative Site, Singapore, Singapore
- South Korea (10):
  - Novartis Investigative Site, Gyeonggi-do, Bucheon Si
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Taiwan (7):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Yilan
- Thailand (4):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Muang

REFERENCES:
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Blood Pressure Drops During Hospitalization for Acute Heart Failure Treated With Serelaxin: A Patient-Level Analysis of 4 Randomized Controlled Trials. Circ Heart Fail. 2022 Apr;15(4):e009199. doi: 10.1161/CIRCHEARTFAILURE.121.009199. Epub 2022 Feb 21. PMID 35184572
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Systolic Blood Pressure and Outcome in Patients Admitted With Acute Heart Failure: An Analysis of Individual Patient Data From 4 Randomized Clinical Trials. J Am Heart Assoc. 2021 Sep 21;10(18):e022288. doi: 10.1161/JAHA.121.022288. Epub 2021 Sep 13. PMID 34514815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * patient randomized : participants who signed ICF (876 participants)
  * Full analyis set: participants who received at least one dose of study drug (870 participants)
  * safety set (858 participtants): participants who received at least one dose of study drug and completed at least one post baseline assessment
Groups:
- Placebo: Patients who received continuous intravenous infusion of matching placebo serelaxin for 48 hours.
- Serelaxin: Patients who receivedcontinuous intravenous infusion of serelaxin for 48 hours.
Period: Overall Study
Arm/Group | Placebo | Serelaxin
Started (876 participants were randomized) | 436 | 440
Full Analysis Set (6 patients were misrandomized and excluded from the fuoll analysis set) | 433 | 437
Safety Set (among these 858 had a least one dose of study drug and at least one post baseline assessment) | 426 | 432
Completed (Phase completion is defined as death or actual follow up greater or equal to Day 165) | 354 | 368
Not Completed | 82 | 72
Not completed — Withdrawal by Subject | 9 | 11
Not completed — study terminated by sponsor | 58 | 54
Not completed — technical problem | 4 | 2
Not completed — patient followd less than 165 days | 11 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set was used
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Serelaxin | Total
Number analyzed (Participants) | 433 | 437 | 870
Age, Continuous [Mean (Standard Deviation); unit: years]
  full analysis set 870 participants | 70.2 (13.86) | 68.9 (14.40) | 69.6 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 147 | 312
  Male | 268 | 290 | 558
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 418 | 420 | 838
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Clinical Composite Endpoint of Treatment Success, Treatment Failure, or no Change.
Description: The trichotomous clinical composite endpoint of treatment success, treatment failure, or no change. Treatment success defined as improvement of dyspnea by Likert scale and at least 2 points improvement by at least 2 physician assessed signs and symptoms (orthopnea, rales edema, and jugular venous pulse) at Day 2; treatment failure defined as worsening heart failure, death, or re-hospitalization due to heart failure or renal failure through Day 5; no change defined as neither the criteria for treatment success nor the criteria for treatment failure was met through Day 5.
Time Frame: through day 5
Population: Full analysis set (FAS) - All patients in the randomized population who were not misrandomized patients. Following the intent-to-treat (ITT) principle, patients were analyzed according to the treatment they had been assigned to at the randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants
  Treatment Failure | 36 | 18
  No Change | 314 | 333
  Treatment Success | 83 | 86

2. Secondary Outcome: Time to WHF
Description: Results are given in terms of number of participants with at least one worsening heart failure (WHF) event through day 5 (pre-defined timeframe).
Time Frame: Through Day 5
Population: Full analysis set (FAS) - All patients in the randomized population who were not misrandomized patients*. Following the intent-to-treat (ITT) principle, patients were analyzed according to the treatment they had been assigned to at the randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants | 26 | 11

3. Secondary Outcome: Time to CV Death
Description: analysis of time to CEC CV death through day 180 : results are given in terms of number of participants with CV death event through day 180 (pre-defined timeframe).
Time Frame: Through Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants | 27 | 27

4. Secondary Outcome: Time to All-cause Death
Description: Results are given in terms of number of participants with all cause death event through day 180 (pre-defined timeframe).
Time Frame: Through Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants | 41 | 33

5. Secondary Outcome: Time to Moderate or Marked Improvements in Dyspnea by Likert Scale, Expressed in Days
Description: Time to event is computed as the number of days from randomization to moderate or marked improvements in dyspnea by Likert scale
Time Frame: Through Day 5
Population: Full analysis set (FAS)with measure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 423 | 429
days | 1.327 (1.4418) | 1.352 (1.5071)

6. Secondary Outcome: Dyspnea by VAS-AUC Changes
Description: Change from baseline in Dyspena by VAS-AUC through Day 5, expressed in mm-hours
Time Frame: Through Day 5
Population: full analysis set with measure
Measure: Mean (Standard Deviation); unit: mm-hours
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 429 | 432
mm-hours | 2284.6 (2702.34) | 2358.2 (2321.17)

7. Secondary Outcome: Length of Intensive Care Unit (ICU) and/or Coronary Care Unit (CCU) Stay for the Index AHF Hospitalization
Description: Length of stay will be defined as the hospitalization discharge date and the time minus the baseline date and time plus 1 day
Time Frame: Up to day 30
Population: full analysis set with measure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 432 | 437
days | 3.2 (5.13) | 2.5 (4.26)

8. Secondary Outcome: Renal Dysfunction and Prevention of Worsening of Renal Function
Description: number of participants with renal dysfunction or in-hospital worsening of renal function through Day 5
Time Frame: Through Day 5
Population: Full analysis set with measure
Measure: Number; unit: participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 418 | 416
participants | 120 | 59

9. Secondary Outcome: Time to Re-hospitalization Due to Heart Failure and Renal Impairment
Description: Time to event is computed as the number of days from randomization to re-hospitalization due to Heart Failure and renal impairment
Time Frame: Through Day 180
Measure: Number; unit: days
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 82
days | 87 | 82

10. Secondary Outcome: Time to CV Death or Re-hospitalization Due to Heart Failure/ Renal Failure
Description: Results are given in terms of number of participants with CV death or at least one re-hospitalization due to Heart Failure through day 180 (pre-defined timeframe).
Time Frame: Through Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants | 87 | 82

11. Secondary Outcome: Time to In-hospital Worsening Heart Failure Through Day 5
Description: Results are given in terms of number of participants with at least one in-hospital worsening heart failure through day 5 (pre-defined timeframe). In-hospital worsening heart failure is defined by symptoms only, signs only, and both symptoms and signs.
Time Frame: Through Day 5
Population: Full analysis set with measure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants
  WHF through day 5 by symptoms | 2 | 1
  WHF through day 5 by signs | 3 | 0
  WHF through day 5 by both | 20 | 9
  death through day 5 | 1 | 1

12. Secondary Outcome: Use of Loop Diuretic and Vasoactive Agents
Description: Number of patients reported with use of loop diuretic and vasoactive agents from randomization through Day 5
Time Frame: Through Day 5
Population: full analysis set with measure
Measure: Number; unit: participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 432 | 437
participants | 58 | 49

13. Secondary Outcome: Change From Baseline in Cardio-renal Biomarkers
Time Frame: Day 2 and Day 5
Population: The data was not collected, and analysis not performed, as the trial was terminated prematurely
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Patients Reported With Total Adverse Events, Serious Adverse Events and Death.
Description: To evaluate the safety and tolerability of intravenous serelaxin in AHF patients, number of patients with total adverse events, serious adverse events and death will be analyzed.
Time Frame: For the safety evaluation, all adverse events will be collected from signing of the informed consent form through Day 5 for non-serious AEs and through Day 14 for serious AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serelaxin
Number analyzed (Participants) | 433 | 437
Participants
  number of participants with SAE | 50 | 37
  number of participants with AE | 253 | 219
  number of patients with death | 41 | 34

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years
Description: AE additional description
Groups:
- RLX030: RLX030
- Total: Total
Arm/Group | RLX030 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 34/432 | 41/426 | 75/858
Serious Adverse Events (participants affected / at risk) | 37/432 | 50/426 | 87/858
Other Adverse Events (participants affected / at risk) | 65/432 | 82/426 | 147/858
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030 (N=432) | Placebo (N=426) | Total (N=858)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 6 | 9
Cardiac failure acute (Cardiac disorders) | 0 | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 2
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 1
Infusion site thrombosis (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Sudden cardiac death (General disorders) | 1 | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Medical device site infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 7 | 13
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Serratia sepsis (Infections and infestations) | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 2 | 1 | 3
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 2
Partial seizures (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 6
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 3 | 3
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 2 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030 (N=432) | Placebo (N=426) | Total (N=858)
Cardiac failure (Cardiac disorders) | 14 | 22 | 36
Constipation (Gastrointestinal disorders) | 23 | 30 | 53
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 39 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However Novartis does not prohibit any inverstigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02007720/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT02007720/SAP_001.pdf